CLINICAL TRIAL: NCT05791071
Title: A Randomized Controlled Phase II Study to Assess the Efficacy of Floreo VR Building Social Connections vs. Active VR Exposure Control as Treatment for Social Skills in Autistic Children
Brief Title: Virtual Reality Intervention for Skill Acquisition Support in Autism Spectrum Disorder (ASD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Floreo, Inc. (Industry)
Collaborators: Cortica (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Floreo Cortica Protocol
Record Dates: First submitted 2023-02-27; First posted 2023-03-30 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Autism Spectrum Disorder
Keywords: ASD; Virtual Reality; VR; Social Communication; Applied Behavior Analysis Therapy
MeSH Terms: conditions — Autism Spectrum Disorder; Communication

STUDY DESIGN:
Intervention Model Description: The two parallel groups include an experimental group that will receive the Floreo VR Building Social Connections program and a control group that will receive non-interventional active VR programing.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects and their parents/caregivers will be blinded to whether they are receiving Floreo VR therapy vs active VR exposure control. Research staff administering the therapy or control will not be blinded to the therapy; however, the clinicians doing pre/post assessments will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Floreo VR Building Social Connections (Experimental): Participants will receive Floreo VR Building Social Connections lessons approximately 3 times a week for no more than 15 minutes per session.
  Interventions: Device: Floreo VR Building Social Connections
- Sham (Sham Comparator): Participants will receive non-interventional active VR videos approximately 3 times a week for no more than 15 minutes per session.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Floreo VR Building Social Connections — Floreo's VR platform consists of a VR headset and wireless tethered VR screens (iPhones) and tablets (iPads) that are seamlessly linked in real time, allowing the therapist (or monitor) to set up lessons, change the interactive environment, and provide live verbal and VR-based guidance, feedback, and rewards to users. The lessons that will be implemented in this intervention are aimed at targeting social skills such as communication, joint attention, and social interactions.
  Arms: Floreo VR Building Social Connections
Device: Sham — This condition will contain the same VR headset and wireless tethered VR screens (iPhones) and tablets (iPads) as the intervention condition, but instead of social skill lessons, only non-intervention, active VR videos such as underwater fish swimming will be shown.
  Arms: Sham

SUMMARY:
A Randomized Controlled Phase II study to assess the efficacy of Floreo VR (Virtual reality) Building Social Connections as treatment for social skills in children with Autism Spectrum Disorder (ASD)

DETAILED DESCRIPTION:
In this randomized controlled phase II study, 30 eligible subjects aged 4-10 years old with documented ASD diagnoses will be enrolled and randomized in a 1:1 ratio intervention vs control group.

The Floreo VR Building Social Connections intervention is designed to be administered for 12 weeks, with three treatment visits per week, for a total of 36 treatment visits.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 4 years to 10 years 11 months of age (up to 11th birthday at randomization).
* Patients or legally authorized representatives must provide written informed consent and be willing and able to comply with study procedures. Participants must provide informed assent as clinically appropriate.
* A diagnosis of autism spectrum disorder on the basis of the clinical judgement of a qualified clinician according to DSM-5 criteria, supported by either the Autism Diagnostic Observation Schedule or the Autism Diagnostic Interview-Revised.
* Participants must receive ABA therapy at Cortica, with scheduled ABA sessions in clinic at least 3 times per week.
* Participants must be able to tolerate VR therapy in the judgement of parent or caregiver and study staff

Exclusion Criteria:

* A history of photosensitive epilepsy, or photoparoxysmal response on electroencephalogram (EEG)
* Active diagnosis of migraine headache or migraine variant (abdominal migraine, cyclic vomiting syndrome), not adequately controlled
* History of balance disorder including vertigo, motion sensitivity, or balance disorder
* Primary sensory impairment (blindness, deafness)
* Motor disorder that would interfere with VR engagement

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Autism Impact Measure (AIM) Assessment | The AIM takes approximately 30 minutes to complete.
  The AIM is a 25-item parent questionnaire targeting sensitivity to change of core ASD symptoms. The questionnaire uses a 2-week recall period with items rated on two corresponding 5-point scales (frequency and impact). The items cover distinct sub-domains of ASD symptoms including Repetitive Behavior, Atypical Behavior, Social Reciprocity, and Peer Interaction. A composite score is also calculated.

SECONDARY OUTCOMES:
CARS-2 | The CARS-3 takes approximately 5-10 minutes to complete after the information needed to make the ratings is collected
  The CARS-2 is a 15-item rating scale used to identify children with autism and determine overall symptom severity. The scale is completed by a clinician familiar with the assessment of ASD after collecting information by direct interview and observation. The rater will also make use of supplemental collected using an unscored Parent/Caregiver Questionnaire. Only the CARS-2 Standard rating scale will be used for the purposes of this study.

OTHER OUTCOMES:
AIM sub-domain scores | The AIM takes approximately 30 minutes to complete.
  The AIM is a 25-item parent questionnaire targeting sensitivity to change of core ASD symptoms. The questionnaire uses a 2-week recall period with items rated on two corresponding 5-point scales (frequency and impact). The items cover distinct sub-domains of ASD symptoms including Repetitive Behavior, Atypical Behavior, Social Reciprocity, and Peer Interaction. A composite score is also calculated.
Vineland-3 Adaptive Behavior Composite and sub-domain scores | The Vineland-3 Comprehensive Interview Form takes approximately 60-90 minutes to complete
  The Vineland-3 evaluates adaptive behavior in five different domains: Social, Communication, Daily Living Skills, and Motor. In the context of this study, it will be administered using the Comprehensive Interview Form, for which a parent or caregiver is interviewed by a qualified rater familiar with the instrument. Based on the summarized scores in each domain, an Adaptive Behavior Composite (ABC) is also calculated. Items are scored on a scale of 0 (never), 1 (sometimes), or 2 (usually) for the level at which the child can independently perform a skill.
Adverse events related to VR use | 5-10 minutes as needed to fill out AE form
  Parents or caregivers will be asked about adverse events at the baseline visit (if this is separate from the screening visit), interim visits 1 and 2, and at the end of study visit. The occurrence or absence of AEs, and a description of any AEs, will be recorded on an Adverse Events Form.

CONTACTS AND LOCATIONS:
Locations (1):
- Cortica, Thousand Oaks, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kanne SM, Mazurek MO, Sikora D, Bellando J, Branum-Martin L, Handen B, Katz T, Freedman B, Powell MP, Warren Z. The Autism Impact Measure (AIM): initial development of a new tool for treatment outcome measurement. J Autism Dev Disord. 2014 Jan;44(1):168-79. doi: 10.1007/s10803-013-1862-3. PMID 23748386
- See also: Floreo Website — http://floreotech.com
- See also: Cortica Website — http://corticacare.com